CLINICAL TRIAL: NCT02361762
Title: Electrophysiological Response to Executive Control Training
Brief Title: Gaming for Autism to Mold Executive Skills Project
Acronym: GAMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Susan Faja, Research Associate, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P00014188; R00HD071966 (NIH)
Record Dates: First submitted 2015-02-04; First posted 2015-02-12 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Autism Spectrum Disorders
Keywords: Executive Function; Theory of Mind; Individual Differences; Social Skills; Executive Control
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Experimental): Computerized executive control training
  Interventions: Behavioral: Computerized executive control training
- Waitlist (No Intervention): The waitlist group will not initially receive the training program. At the end of the study, the waitlist group will be offered training if it is efficacious.

INTERVENTIONS:
Behavioral: Computerized executive control training — Children will play computerized training games designed to improve executive control skills. Each training activity is structured to achieve a particular type of training related to executive control and/or attention shifting.
  Sessions last for 1 hour each and the intensity of intervention ranges from 5-10 hours. Children will receive training until all levels of all tasks have been passed or 10 hours, whichever happens first. All training exercises have a number of levels, and children progress to the next level by meeting specific criteria for accuracy and/or speed.
  A trainer will be present during all sessions to help children comply with the training demands and to teach skills involved in completing challenging tasks.
  Arms: Training

SUMMARY:
The goal of the project is to better understand executive control-how children manage complex or conflicting information in the service of a goal. This skill has been linked to social and academic functioning in typically developing children. Executive control is often reduced in children with autism spectrum disorder (ASD), but it has not been a focus of treatment. This project will have the goal of determining whether computer-training tasks developed to enhance the executive control skills of preschoolers and school-aged children without autism are appropriate for children with ASD. The investigators do not yet know if this training is beneficial for children with ASD. In addition, because executive control has been found to relate to social knowledge and problem solving, the investigators will collect information with this type of task to measure possible effects of training.

DETAILED DESCRIPTION:
Participation will include two phone calls to determine if the study is a good fit and collect some preliminary information, five visits to Boston Children's Hospital (3 before training and 2 about 6-8 weeks later), caregiver questionnaires, and an optional teacher questionnaire packet. The visits will include activities designed to assess verbal and nonverbal thinking ability; social skills and general interests; and specific tasks related to cognitive and social problem solving. In addition, EEG measurement of brain function will be made. EEG is a non-invasive recording of brain activity. Children will be randomly assigned (i.e., like flipping a coin) to receive training or to a non-training group. The training group will complete tasks designed to improve executive control presented over the course of 5-10 1-hour sessions. All tasks are game-like and are presented on a computer with child friendly graphics. A staff member will work with each child as he/she completes the training activities. Children assigned to the non-training group will be invited to participate in training at the end of the study if it is shown to improve executive control.

ELIGIBILITY:
Inclusion Criteria:

* Children should be 7 to 11 years of age
* Children must have a parent/guardian who is available and willing to provide informed consent and to respond to screening phone calls
* Children should have an existing diagnosis of an autism spectrum disorder, which will be confirmed using research measures and criteria
* Children must have general cognitive ability in the average range or above (above 80 using the Wechsler Abbreviated Scale of Intelligence-2 Full Scale IQ)
* Caregivers and children must be fluent in English

Exclusion Criteria:

* Children must not have a seizure disorder or be taking medication that alters EEG processes (e.g. anti-seizure medications)
* Children must not have medical disorders or injuries affecting the brain or spinal cord
* Children may not have experienced significant prenatal exposure to substances such as tobacco, alcohol or street drugs
* Children may not have significant sensory or motor impairment that would limit the ability to participate in table top or EEG testing, or make responding during computer activities difficult

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Faja, Ph.D., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital: Labs of Cognitive Neuroscience- Faja Lab, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Edmunds SR, MacNaughton GA, Rueda MR, Combita LM, Faja S. Beyond group differences: Exploring the preliminary signals of target engagement of an executive function training for autistic children. Autism Res. 2022 Jul;15(7):1261-1273. doi: 10.1002/aur.2735. Epub 2022 Apr 28. PMID 35481725
- See also: Faja Lab Website — http://www.childrenshospital.org/research-and-innovation/research/labs/faja-laboratory

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, 106 potential participants were screened. 31 were ineligible; 5 others declined to participate.
  70 children were randomized. 35 were assigned to training. 35 were assigned to waitlist.
Groups:
- Training: Computerized executive control training
  Computerized executive control training: Children will play computerized training games designed to improve executive control skills. Each training activity is structured to achieve a particular type of training related to executive control and/or attention shifting.
  Sessions last for 1 hour each and the intensity of intervention ranges from 5-10 hours. Children will receive training until all levels of all tasks have been passed or 10 hours, whichever happens first. All training exercises have a number of levels, and children progress to the next level by meeting specific criteria for accuracy and/or speed.
  A trainer will be present during all sessions to help children comply with the training demands and to teach skills involved in completing challenging tasks.
Period: Overall Study
Arm/Group | Training | Waitlist
Started | 35 | 35
Completed | 35 | 33
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Training | Waitlist | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.80 (1.39) | 8.69 (1.41) | 8.704 (1.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 32 | 31 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 31 | 34 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 29 | 27 | 56
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change Task - Stop Signal Reaction Time
Description: Conflict Processing-Behavior (Post-testing controlling for Baseline) Children indicate the location of a picture by pressing the left and right arrow buttons for 75% of the trials (i.e., the dominant task).
  For the remaining 25% of trials, a stop signal appears and a Change response (i.e., space bar) was required. Stop signals occurred equally at 50, 200, 350, and 500 ms before the anticipated response based on the child's reaction time.
  The SSRT estimates the latency of inhibitory responding to the stop signal. Lower scores indicate more rapid inhibition.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Of the 68 children randomized who returned for post testing, data were available for 61 across both time points; one participant was unable to map the correct buttons at baseline, two participants refused the task at post testing, and computer failure occurred for four participants (3 at baseline, 1 at post testing).
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 31 | 30
miliseconds
  Baseline | 233.8 (87.8) | 238.3 (94.3)
  Post-training/Waitlisted phase | 213.6 (78.5) | 234.7 (98.1)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.36, ANCOVA; ANCOVA-of-change was used to compare the Training and Waitlist groups at post-testing while controlling for baseline (baseline was co-varied)

2. Primary Outcome: Stroop Task (Difference in Percentage of Correct Responses for Congruent Minus Incongruent Trials)
Description: Conflict Processing-Behavior (Post-testing controlling for Baseline) Trials were presented in three conditions: (1) congruent trials (25%); (2) incongruent trials (25%); and (3) neutral trials (50%). The difference between percent correct for congruent and incongruent conditions was the dependent variable, such that larger differences indicated more difficulty with conflicting information. Lower scores at Post-testing indicate improved ability to suppress interfering/conflicting information.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Data were available for 63 children; five children were unable to complete the task or refused to play (3 baseline, 2 at post).
Measure: Mean (Standard Deviation); unit: difference in % of correct responses
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 34 | 29
difference in % of correct responses
  Baseline | 3.8 (8) | 6.0 (12)
  Post-Training/Wait-listed phase | 2.9 (13) | 3.8 (9)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.79, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Event-related Potentials Assessed During Child Attention Network Flanker Task
Description: Conflict Processing-Event Related Potential (ERP) Brain Response (N2 mean amplitude) Data were compared for congruent and incongruent conditions at each time point (baseline and post testing).
  Each trial of the task began with a beep for 150ms paired with a fixation cross for 450ms at the center of the screen. Then, a target and flankers were presented for 2000ms. Congruent trials (50%) consisted of a central target animal flanked by two animals on each side with the same orientation and size as the target. Incongruent trials (50%) were identical except that the target and flankers faced opposite directions. Children pressed a button indicating the direction the target animal faced (50% left, 50% right) and received visual and auditory feedback upon responding.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 24 | 22
microvolts
  Congruent - Pre | -.20 (3.2) | -2.5 (3.3)
  Incongruent - Pre | .83 (3.3) | -3.8 (4.8)
  Congruent - Post | -1.0 (3.6) | -3.7 (4.1)
  Incongruent - Post | -1.8 (3.7) | -3.3 (4.5)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.009, ANOVA; Repeated measures ANOVA compared group (Training/Waitlist) by time (Pre/Post) by condition (Congruent/Incongruent)

4. Primary Outcome: BRIEF Parent Survey (Global Executive Composite)
Description: Executive Control at home/school-Generalization (Post-testing controlling for Baseline) Global Executive Composite (GEC) scores are available for parents. The GEC is comprised of two sub-scales: Metacognition and Behavioral Regulation.
  T-scores are reported for the GEC (range = 30-100). Higher scores reflect more difficulty with executive function. At Post, lower scores represent a better outcome.
  Note: Teacher BRIEF was originally planned as an outcome measure, but due to low teacher response (10 teachers provided data for each group at both time points) the results were not analyzed.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: 63 parents completed the questionnaire at both time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 33 | 30
scores on a scale
  Global Executive Composite-Pre | 66.55 (11.51) | 68.40 (8.61)
  Global Executive Composite-Post | 65.85 (9.96) | 67.77 (10.42)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = .79, ANCOVA — ANCOVA-of-change was used to compare the Training and Waitlist groups at post-testing while controlling for baseline (baseline was co-varied); Compared scores at post testing with baseline scores covaried

5. Secondary Outcome: Backward Digit Span (Scaled Score)
Description: Working Memory Behavior (Post-testing controlling for Baseline) A control task - not specifically targeted by intervention. Scaled score for Backward Digit Span (higher scores represent better memory).
  Scaled scores are reported (range = 1-19). Higher scores reflect better working memory (an aspect of executive function). At Post, higher scores represent a better outcome.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Of the 68 children who completed post testing, 63 provided data at both time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 33 | 30
scores on a scale
  Baseline | 10.42 (3.45) | 9.83 (3.55)
  Post-training/Waitlisted phase | 10.15 (3.17) | 9.55 (3.55)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.61, ANCOVA; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Social Attribution Task (SAT) - Problem Solving Scale
Description: Theory of Mind Behavior (Post-testing controlling for Baseline) A measure of generalization.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Of the 68 children who returned for post testing, 45 children had sufficient time during visits at both time points for this task.
Measure: Mean (Standard Deviation); unit: percent correct on SAT problem solving
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 24 | 21
percent correct on SAT problem solving
  Baseline | 34.6 (16.4) | 33.8 (16.9)
  Post-Training | 32.9 (16.3) | 31.0 (15.1)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.68, ANCOVA; ANCOVA-of-change was used to compare the Training and Waitlist groups at post-testing while controlling for baseline (baseline was co-varied)0

7. Secondary Outcome: Theory of Mind Composite: Perception Knowledge, Location Change False Belief, Unexpected-contents False Belief
Description: Theory of Mind (TOM) Behavior (Post-testing controlling for Baseline) A measure of generalization Composite score by computing the percent correct (range = 0-100% correct) across three video tasks measuring cognitive aspects of theory of mind (i.e., the Perception Knowledge Task, Location Change False Belief Task, and Unexpected-contents False Belief Task). Higher scores represent better performance (i.e., more correct responses). Higher scores at post testing represent better outcomes.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Of the 68 children who returned for post testing, 60 children had sufficient time during visits at both time points to complete these video tasks.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 31 | 29
percentage of correct responses
  Baseline | 75 (25) | 71 (29)
  Post-training/Waitlisted phase | 90 (20) | 84 (26)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.54, ANCOVA; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: TOM Test (Theory of Mind Test)
Description: Theory of Mind Behavior (Post-testing controlling for Baseline). A measure of generalization. Overall percent correct across the three sub-scales (i.e., percent correct calculated across all items of Level 1-Precursors, Level 2-First Order False Belief, and Level 3-Advanced) is reported. The percent correct ranges from 0-100% correct. Higher scores represent better theory of mind (affective and first/second order false belief).
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Of the 68 children who returned for post testing, 67 had sufficient time to complete the TOM Test at both time points.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 34 | 33
percentage of correct responses
  Baseline | 66 (14) | 63 (13)
  Post-Training/Wait-listed phase | 71 (12) | 65 (10)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.08, ANCOVA; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Social Skills Improvement System-Parent (SSIS) - Social Standard Score
Description: Social function home (Post-testing controlling for Baseline). A measure of generalization. Scores were available from parents. The SSIS Social Scale organizes prosocial behaviors into seven areas or subscales: Communication, Cooperation, Assertion, Responsibility, Empathy, Engagement, and Self-Control. Scores range from 40-160. Higher scores reflect more prosocial skills (i.e., better social ability). At Post, higher scores represent a better outcome.
  Note: Teacher SSIS was originally planned as an outcome measure, but due to low teacher response the results were not analyzed.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Of the 68 children who returned for post testing, 62 parents completed the SSIS questionnaire at both time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 32 | 30
scores on a scale
  Baseline | 81.63 (12.5) | 80.47 (15.7)
  Post-training/Waitlisted phase | 81.69 (10.6) | 79.33 (14.2)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.37, ANCOVA; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Narrative Language Task
Description: Social Communication Ability Behavior (Post-testing controlling for Baseline). A measure of generalization.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Data were not collected.
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Performance on Hungry Donkey Task Assessed as Ratio of Safe to Risky Selections
Description: Conflict Processing (Reward) Behavior (Post-testing controlling for Baseline). Children selected from four doors with varying reward and loss ratios. Two doors have lower rewards but an overall net gain (safe) and two doors have higher rewards but an overall net loss (risky). Scores represent the ratio of safe to risky selections in the final two blocks (of five total blocks administered).
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Of the 68 children who completed post-testing, 64 completed the task at both time points.
Measure: Mean (Standard Deviation); unit: ratio of safe to risky selections
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 33 | 31
ratio of safe to risky selections
  Baseline | 1.39 (10.85) | 0.16 (10.28)
  Post-training/Waitlisted phase | 0.33 (11.7) | 1.74 (11.9)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.62, ANCOVA; [statistical method as in outcome 1, analysis 1]

12. Secondary Outcome: Event-related Potentials Assessed During Cued Go/Nogo Task
Description: Conflict Processing-ERP Brain Response (N2 mean amplitude) Data were compared for Go and Nogo conditions at each time point (baseline and post testing).
  The task included 200 test trials. During 'go' trials (70% of trials), children were instructed to press a single button on a keypad each time a letter appeared on the screen. During 'nogo' trials (30% of trials), children were instructed to withhold their response when a specific letter appeared on the screen. To account for the confound of frequency with condition, two letters were used for go trials - an infrequent go (30% of trials) and a frequent go (40% of trials). Go responses were analyzed only for the infrequent go trials. Each trial was preceded by a fixation cross presented on the screen for 500 ms. Test trials were then presented for 700 ms. Only ERPs for correct trials that followed a correct 'go' response were analyzed in order to ensure consistent motor response on the previous trial.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: This task was always administered after the Child ANT Flanker Task, resulting in fewer children who completed it at both time points. Of the 68 children who returned for post-testing, 31 provided usable, artifact free data at both time points.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 16 | 15
microvolts
  Go - Pre | -2.4 (2.8) | -2.9 (4.0)
  Nogo - Pre | -1.6 (3.4) | -3.0 (4.3)
  Go - Post | -1.1 (2.1) | -2.3 (3.0)
  Nogo - Post | -2.8 (3.6) | -2.6 (4.5)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.10, ANCOVA; Repeated measures ANOVA compared group (Training/Waitlist) by time (Pre/Post) by condition (Go/Nogo)

13. Post Hoc Outcome: Repetitive Behavior Scale-Revised (RBS-R) - Total Score
Description: Parent report of restricted and repetitive symptoms at home-Generalization (Post-testing controlling for Baseline) Total RBS-R scores are analyzed. The RBS-R includes information about stereotyped behavior, self-injurious behavior, compulsive behavior, ritualistic behavior, sameness behavior, and restricted behavior. The range of scores is (range = 0-176). Higher scores reflect more restricted and repetitive behavior symptoms. At Post, lower scores represent a better outcome.
Time Frame: Baseline (Pre Training/Waitlist Phase) and at 11-12 Weeks (Post Training/Waitlist Phase)
Population: Of the 68 children who returned for post-testing, data were available for 60 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training | Waitlist
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 16.61 (10.75) | 24.11 (14.06)
  Post-training/Waitlisted phase | 13.61 (9.04) | 27.03 (17.90)
Statistical Analysis 1: Comparison: Training vs Waitlist; Test type: Other; p = 0.02, ANCOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Given that this was a behavioral study, adverse event data were not formally collected but participants were encouraged to report any concerns about participation to study staff throughout the study period, which was approximately 6 months (baseline + 3 month intervention window + post testing). At each assessment visit, families were also given a debriefing form to determine whether the child's behavior was expected during the visit and whether any stressors occurred since the previous visit.
Arm/Group | Training | Waitlist
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT02361762/Prot_SAP_000.pdf